CLINICAL TRIAL: NCT03194633
Title: Effectiveness and Tolerability of Long-Acting Nifedipine Gastrointestinal Therapeutic System in Chronic Kidney Disease With Uncontrolled Hypertension Patients, a Prospective, Multicenter, Observational Study
Acronym: ADRENAL
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 18679
Record Dates: First submitted 2017-06-20; First posted 2017-06-21 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Nifedipine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nifedipine controlled-release tablets(Nifedipine GITS, ADALAT, BAYA1040): Male and female patients with a diagnosis of CKD and hypertension (age, 18-70 years) was enrolled.
  Interventions: Drug: Nifedipine controlled-release tablets(Nifedipine GITS, ADALAT, BAYA1040)

INTERVENTIONS:
Drug: Nifedipine controlled-release tablets(Nifedipine GITS, ADALAT, BAYA1040) — Nifedipine GITS 60 mg (once per day)

SUMMARY:
Chronic kidney disease (CKD) and hypertension are two closely related common chronic diseases that have serious implications to human health. Hypertension is a major cause for progression of renal disease and a risk factor for cardiovascular disease (CVD). Control of Blood Pressure (BP) to target is now considered to be the main goal in the treatment of patients with CKD.

In clinical practice, it is difficult for CKD patients with hypertension to achieve systolic BP (SBP) or diastolic BP (DBP) goal; oftentimes, calcium channel blocker (CCB) class of drugs, for example, nifedipine gastrointestinal therapeutic system (GITS), is used in such patients. Previous data have demonstrated nifedipine to be having a significant dose-response relationship; that is, nifedipine 60 mg provided better BP reduction than 30 mg. However, there are limited studies that have evaluated the efficacy and tolerability of nifedipine GITS 60 mg in Chinese CKD patients with hypertension. Hereby, the objective of this study was to evaluate the effectiveness and tolerability of nifedipine GITS 60 mg treatment in a large cohort of CKD patients with uncontrolled hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18-70 years
* Patients diagnosed with CKD (Estimated Glomerular Filtration Rate (eGFR) >15 mL/min/1.73 m*2) and hypertension without dialysis/replacement therapy
* Patients with uncontrolled hypertension (office SBP ≥140 mmHg and DBP ≥ 80 mmHg) who have received Renin-Angiotensin System Inhibitors (RASI) treatment or have not received RASI treatment because of any contraindications
* Patients who haven't received nifedipine GITS 60 mg (once per day) previously
* Patients for whom the decision to initiate treatment with nifedipine GITS 60 mg was made as per the investigator's routine treatment practice
* Signed informed consent
* No participation in an investigational program with interventions outside of routine clinical practice

Exclusion Criteria:

* Have a contraindication to nifedipine GITS according to the approved prescribing information
* Patients participating in an investigational program with interventions outside of routine clinical practice

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are prescribed 60-mg nifedipine GITS (once per day) and meet the inclusion/exclusion criteria will be enrolled into the study.
Sampling Method: Non-Probability Sample
Enrollment: 871 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2020-05-14 (Actual); Study Completion 2020-08-28 (Actual)

PRIMARY OUTCOMES:
Change in office systolic blood pressure from baseline to week 12 | At week 12
  Change in office systolic blood pressure from baseline to week 12

SECONDARY OUTCOMES:
Change in office diastolic blood pressure from baseline to week 12 | At week 12
  Change in office diastolic blood pressure from baseline to week 12
Change in systolic blood pressure and diastolic blood pressure from baseline to week 12 according to baseline SBP stratification | At week 12
  Change in systolic blood pressure and diastolic blood pressure from baseline to week 12 according to baseline SBP stratification, stratified by two subgroups baseline, SBP 140-160 mmHg and ≥ 160 mmHg
Change in systolic blood pressure and diastolic blood pressure from baseline to week 12 at different stages of Chronic Kidney Disease | At week 12
  Change in systolic blood pressure and diastolic blood pressure from baseline to week 12 at different stages of Chronic Kidney Disease, stage 1 to stage 5
Systolic blood pressure and diastolic blood pressure control rate at week 12 | At week 12
  Systolic blood pressure and diastolic blood pressure control rate at week 12
Number of participants with adverse events and serious adverse events | At week 12

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Multiple Locations, China

REFERENCES:
- [Derived] Lv R, Chen J, Wang H, Wang J, Cheng H, Li R, Li W, Zhang T, Wei L, Chen Q, Huang J, Yu F, Shen S, Wu H, Liu C, Hong F, Liu J, Zhang X, Xiao H, Song W. Effectiveness and Tolerability of Nifedipine GITS in Patients with Chronic Kidney Disease and Uncontrolled Hypertension: A Prospective, Multicenter, Observational Study (ADRENAL). Adv Ther. 2021 Sep;38(9):4771-4785. doi: 10.1007/s12325-021-01850-3. Epub 2021 Jul 30. PMID 34331258